CLINICAL TRIAL: NCT05486429
Title: Evaluation of Lipid Profile in Different Grades of Non-alcoholic Fatty Liver Disease Diagnosed by Ultrasound
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Nashwa Khalaf Refaie, Resident at Tropical Medicine and Gastroenterology, Sohag University
Other Study IDs: Soh-med-22-07-18
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Combination Product: Abdominal ultrasound and lipid profile — All patients will be subjected to: -
  * Complete history taking with stress on:
    * Age, sex, comorbid conditions (diabetes, hypertension, ischemic heart disease)
    * History of intake of lipid lowering drugs.
  * Thorough clinical examination:
  General examination, vital sign, height, weight, body mass index. Abdominal examination (hepatomegaly, splenomegaly, ascites)
  * Laboratory Investigation:
    1.Lipid profile (total cholesterol, triglyceride, HDL, LDL, VLDL (
    .2Liver function tests (ALT, AST, Albumin, Bilirubin, PT, PC, INR) 3.Complete blood picture. 4.Serology for HBV, HCV. 5.Serum creatinine. 6.Fasting and postprandial blood sugar.
  * Radiological Investigation:
    1.Abdominal ultrasound.
  * FIB - 4 it combines platelets count, ALI, AST and age.
  * AST/Platelets ratio index is calculated as (AST/upper limit of normal range) /Platelets count (10^9/L) ×100.

SUMMARY:
Liver cells play a major role in the regulation of lipid metabolism. They are the principal location for lipoprotein and cholesterol synthesis. In healthy individuals an equilibrium is preserved between utilization, biosynthesis and transfer of lipid fractions. Many diseases that affect the parenchyma of liver can lead to changes in the structure of lipoprotein and transport through blood.

Non - alcoholic fatty liver disease (NAFLD) is an abnormal accumulation of fat in the liver in the absence of secondary causes of fatty liver, such as significant alcohol use, viral hepatitis or medications that induce fatty liver. NAFLD is the most common liver disorder worldwide and is present in approximately 25%of the world's population [3].

People with NAFLD often have no symptoms and NAFLD is often only detectable during routine blood tests or unrelated abdominal imaging or liver biopsy [4].in some cases NAFLD can cause symptoms such as fatigue, malaise and dull right upper quadrant abdominal discomfort. Non - alcoholic steatohepatitis can severely impair liver functions leading to cirrhosis, liver failure and hepatocellular carcinoma.

Grading of NAFLD on ultrasound: when the echogenicity is only marginally increases, it is grade 1, when the echogenic liver obscures the echogenic walls of portal vein branches, it is grade 2, and when the echogenic liver obscures the diaphragmatic outlines, it is grade 3 fatty infiltrations.

DETAILED DESCRIPTION:
Liver cells play a major role in the regulation of lipid metabolism. They are the principal location for lipoprotein and cholesterol synthesis. In healthy individuals an equilibrium is preserved between utilization, biosynthesis and transfer of lipid fractions. Many diseases that affect the parenchyma of liver can lead to changes in the structure of lipoprotein and transport through blood.

Non - alcoholic fatty liver disease (NAFLD) is an abnormal accumulation of fat in the liver in the absence of secondary causes of fatty liver, such as significant alcohol use, viral hepatitis or medications that induce fatty liver [3]. NAFLD is the most common liver disorder worldwide and is present in approximately 25%of the world's population.

People with NAFLD often have no symptoms and NAFLD is often only detectable during routine blood tests or unrelated abdominal imaging or liver biopsy.in some cases NAFLD can cause symptoms such as fatigue, malaise and dull right upper quadrant abdominal discomfort [5]. Non - alcoholic steatohepatitis can severely impair liver functions leading to cirrhosis, liver failure and hepatocellular carcinoma.

Grading of NAFLD on ultrasound: when the echogenicity is only marginally increases, it is grade 1, when the echogenic liver obscures the echogenic walls of portal vein branches, it is grade 2, and when the echogenic liver obscures the diaphragmatic outlines, it is grade 3 fatty infiltrations.

Liver biopsy is a sensitive method for diagnosis of NAFLD. However, liver biopsy is painful and invasive procedure with rare, but potentially life-threatening complications like bleeding and is prone to sampling error.

Circulating serum biomarkers of liver fibrosis can give moderate estimates in the diagnosis of liver fibrosis and cirrhosis. The ratio of AST to platelets known as AST /Platelets ratio index (APRI Score) and Fibrotest are recommended as the preferred non invasive tests for cirrhosis by the Asian -Pacific Association for Study of the Liver (APASL).Several other scores such as FIB -4 score and NAFLD fibrosis score can also reflect the burden of fibrosis in the liver.

Dyslipidemia: hypertriglyceridemia, low HDL-C level and high LDL-C level is the most frequent type of lipid abnormality in NAFLD. Previous studies demonstrated that decreased HDL-C levels were associated with occurrence of NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who have non - alcoholic fatty liver by ultrasonography (18-65 years old).

Exclusion Criteria:

* HCV, HBV patients.
* Alcoholic patients
* Patients under treatment with lipid lowering drugs.
* Patients under treatment with steatogenic drugs.
* Patients taking hepatotoxic drugs.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will include all adult patients with non - alcoholic fatty liver disease will attend to outpatient clinic of Tropical Medicine Department, Sohag University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-07-20 (Actual); Primary Completion 2023-01-20 (Estimated); Study Completion 2023-01-20 (Estimated)

PRIMARY OUTCOMES:
Lipid profile | 6 months
  serum total cholesterol, triglyceride, HDL, LDL, VLDL

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Marjot T, Moolla A, Cobbold JF, Hodson L, Tomlinson JW. Nonalcoholic Fatty Liver Disease in Adults: Current Concepts in Etiology, Outcomes, and Management. Endocr Rev. 2020 Jan 1;41(1):bnz009. doi: 10.1210/endrev/bnz009. PMID 31629366
- [Background] Chalasani N, Younossi Z, Lavine JE, Charlton M, Cusi K, Rinella M, Harrison SA, Brunt EM, Sanyal AJ. The diagnosis and management of nonalcoholic fatty liver disease: Practice guidance from the American Association for the Study of Liver Diseases. Hepatology. 2018 Jan;67(1):328-357. doi: 10.1002/hep.29367. Epub 2017 Sep 29. No abstract available. PMID 28714183
- [Background] Friedman SL, Neuschwander-Tetri BA, Rinella M, Sanyal AJ. Mechanisms of NAFLD development and therapeutic strategies. Nat Med. 2018 Jul;24(7):908-922. doi: 10.1038/s41591-018-0104-9. Epub 2018 Jul 2. PMID 29967350
- [Background] Peng K, Mo Z, Tian G. Serum Lipid Abnormalities and Nonalcoholic Fatty Liver Disease in Adult Males. Am J Med Sci. 2017 Mar;353(3):236-241. doi: 10.1016/j.amjms.2017.01.002. Epub 2017 Jan 11. PMID 28262209